CLINICAL TRIAL: NCT07102862
Title: Unveiling Altered Hemorheology in Adolescent Idiopathic Scoliosis: a Cross-sectional Case-control Study
Brief Title: Altered Hemorology in Adolescent Idıopathic Scoliosis
Acronym: AHIAIS
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Aslinur Keles Ercisli, MD, PhD, Principal investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: AHIAIS-2025; SBU-2025 (Other: University of Health Sciences)
Record Dates: First submitted 2025-07-09; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Adolescent Scoliosis
Keywords: Idiopathic Adolescent Scoliosis; hemorheology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 10-18 years old AIS patients
- Control Healthy Subjects: Sex and aged match healthy subjecyts

SUMMARY:
This study aims to investigate potential alterations in hemorheological parameters in adolescents with idiopathic scoliosis (AIS) compared to healthy controls. A total of 30 AIS patients and 30 age- and sex-matched healthy individuals will be evaluated through clinical, radiological, and laboratory assessments. Hematocrit, plasma and whole blood viscosity, erythrocyte deformability, and aggregation will be measured. The goal is to determine whether structural spinal deformities in AIS are associated with changes in microcirculatory blood flow properties.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is the most common type of scoliosis in children and adolescents. Although extensively studied from orthopedic and biomechanical perspectives, its potential systemic effects remain poorly understood. This study is designed to investigate whether AIS is associated with alterations in blood rheology-specifically, changes in viscosity, erythrocyte deformability, and aggregation-which may reflect underlying microcirculatory dysfunction.

Hemorheology refers to the study of blood flow and its mechanical properties. In this study, key hemorheological parameters-including hematocrit (Hct), whole blood viscosity (WBV), plasma viscosity (PV), erythrocyte deformability (ED), and erythrocyte aggregation (EA)-will be assessed in AIS patients and healthy controls. A total of 30 AIS patients and 30 age- and sex-matched healthy participants will be enrolled.

Blood samples will be collected for rheological analysis, and measurements will be performed using a rotational cone-plate viscometer and a laser-optical erythrocyte analyzer under standardized shear conditions. Clinical and radiological data, such as Cobb angle, vertebral rotation, and sagittal alignment, will also be collected. Statistical comparisons between groups and correlation analyses will be conducted to evaluate the relationships between hemorheological variables and scoliosis severity or type.

This study will provide the first controlled assessment of hemorheological behavior in adolescents with idiopathic scoliosis. Results may offer novel insights into whether spinal deformity has systemic circulatory implications and may help identify early markers of microvascular dysfunction associated with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Presence of structural scoliosis with a Cobb angle greater than 10°
* Age between 10 and 18 years

Exclusion Criteria:

* Other types of scoliosis, such as syndromic conditions, congenital vertebral deformities, and neuromuscular scoliosis
* Presence of any diseases or conditions that may affect hemorheology, such as cardiovascular, respiratory, and hematologic diseases
* Obesity (Body mass index [BMI] > 30)
* Being treated surgically for scoliosis

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This case-control study occurred at the University of Health Sciences in Istanbul from January to May 2025. Participation was voluntary, and written informed consent was obtained from both the adolescents and their legal guardians prior to data collection. Adolescents with idiopathic scoliosis will initially be recruited. An equal number of age-matched and sex-matched healthy controls will also be included. All participants will undergo the same evaluation protocol, and inclusion/exclusion criteria will be applied consistently across both groups.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Plasma viscosity (PV) | At baseline (single time point)
  Measurement of plasma viscosity (mPa·s) using cone-plate viscometry at a shear rate of 450 s-¹.
Whole blood viscosity (WBV) | At baseline (single time point)
  Measurement of whole blood viscosity (mPa·s) using cone-plate viscometer at multiple shear rates (37.5 to 450 s-¹).
Erythrocyte deformability (EImax) | At baseline (single time point)
  Evaluation of erythrocyte elongation index (EImax) using laser-assisted ektacytometry (Lorrca MaxSis).
Erythrocyte deformability (SS1/2) | At baseline (single time point)
  Evaluation of shear stress at half EImax (SS1/2) using laser-assisted ektacytometry (Lorrca MaxSis).
Erythrocyte aggregation (AI and Tr) | At baseline (single time point)
  Measurement of aggregation index (AI) using Lorrca MaxSis at 37°C under standardized conditions.
Erythrocyte aggregation (Tr) | At baseline (single time point)
  Measurement of relaxation time (Tr) using Lorrca MaxSis at 37°C under standardized conditions.

SECONDARY OUTCOMES:
Correlation between Cobb angle and the Plasma viscosity (mPa·s) | At baseline (single time point)
  Plasma viscosity (mPa·s), measured using a cone-plate rotational viscometer at 450 s-¹, and Cobb angle measured in degrees on standing posteroanterior spinal radiographs
Correlation between cervical lordosis angle and the Plasma viscosity (mPa·s) | At baseline (single time point)
  Plasma viscosity (mPa·s), measured using a cone-plate rotational viscometer at 450 s-¹, and cervical lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between thoracic kyphosis angle and the Plasma viscosity (mPa·s) | At baseline (single time point)
  Plasma viscosity (mPa·s), measured using a cone-plate rotational viscometer at 450 s-¹, and thoracic kyphosis angle measured in degrees on standing lateral spinal radiographs
Correlation between lumbar lordosis angle and the Plasma viscosity (mPa·s) | At baseline (single time point)
  Plasma viscosity (mPa·s), measured using a cone-plate rotational viscometer at 450 s-¹, and lumbar lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between angle of trunk rotation (ATR) and the Plasma viscosity (mPa·s) | At baseline (single time point)
  Plasma viscosity (mPa·s), measured using a cone-plate rotational viscometer at 450 s-¹, and angle of trunk rotation (ATR) measured with a scoliometer
Correlation between vertebral rotation (Nash-Moe grade) and the Plasma viscosity (mPa·s) | At baseline (single time point)
  Plasma viscosity (mPa·s), measured using a cone-plate rotational viscometer at 450 s-¹, and Vertebral rotation will be assessed using the Nash-Moe grading system on standing posteroanterior spinal radiographs. The Nash-Moe method classifies pedicle asymmetry into 5 grades (Grade 0 to Grade 4), where higher grades indicate increased vertebral rotation.
Correlation between joint hypermobility (Beighton score) and the Plasma viscosity (mPa·s) | At baseline (single time point)
  Plasma viscosity (mPa·s), measured using a cone-plate rotational viscometer at 450 s-¹, and Joint hypermobility will be measured using the Beighton score (0-9 scale), a standardized clinical examination evaluating passive dorsiflexion of the fifth finger, thumb apposition, elbow hyperextension, knee hyperextension, and forward flexion of the trunk. Scores ≥5 will be considered indicative of generalized joint hypermobility.
Correlation between Cobb angle and the Whole blood viscosity (mPa·s) | At baseline (single time point)
  Whole blood viscosity (mPa·s), measured at multiple shear rates (37.5 to 450 s-¹) and Cobb angle measured in degrees on standing posteroanterior spinal radiographs
Correlation between cervical lordosis angle and the Whole blood viscosity (mPa·s) | At baseline (single time point)
  Whole blood viscosity (mPa·s), measured at multiple shear rates (37.5 to 450 s-¹) and cervical lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between thoracic kyphosis angle and the Whole blood viscosity (mPa·s) | At baseline (single time point)
  Whole blood viscosity (mPa·s), measured at multiple shear rates (37.5 to 450 s-¹) and thoracic kyphosis angle measured in degrees on standing lateral spinal radiographs
Correlation between lumbar lordosis angle and the Whole blood viscosity (mPa·s) | At baseline (single time point)
  Whole blood viscosity (mPa·s), measured at multiple shear rates (37.5 to 450 s-¹), and lumbar lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between angle of trunk rotation (ATR) and the Whole blood viscosity (mPa·s) | At baseline (single time point)
  Whole blood viscosity (mPa·s), measured at multiple shear rates (37.5 to 450 s-¹), and angle of trunk rotation (ATR) measured with a scoliometer
Correlation between vertebral rotation (Nash-Moe grade) and the Whole blood viscosity (mPa·s) | At baseline (single time point)
  Whole blood viscosity (mPa·s), measured at multiple shear rates (37.5 to 450 s-¹), and Vertebral rotation will be assessed using the Nash-Moe grading system on standing posteroanterior spinal radiographs. The Nash-Moe method classifies pedicle asymmetry into 5 grades (Grade 0 to Grade 4), where higher grades indicate increased vertebral rotation.
Correlation between joint hypermobility (Beighton score) and the Whole blood viscosity (mPa·s) | At baseline (single time point)
  Whole blood viscosity (mPa·s), measured at multiple shear rates (37.5 to 450 s-¹), and Joint hypermobility will be measured using the Beighton score (0-9 scale), a standardized clinical examination evaluating passive dorsiflexion of the fifth finger, thumb apposition, elbow hyperextension, knee hyperextension, and forward flexion of the trunk. Scores ≥5 will be considered indicative of generalized joint hypermobility.
Correlation between Cobb angle and Erythrocyte deformability (EImax) | At baseline (single time point)
  Erythrocyte deformability (EImax), measured using laser-optical ektacytometry (Lorrca MaxSis) and Cobb angle measured in degrees on standing posteroanterior spinal radiographs
Correlation between cervical lordosis angle and Erythrocyte deformability (EImax) | At baseline (single time point)
  Erythrocyte deformability (EImax), measured using laser-optical ektacytometry (Lorrca MaxSis) and cervical lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between thoracic kyphosis angle and Erythrocyte deformability (EImax) | At baseline (single time point)
  Erythrocyte deformability (EImax), measured using laser-optical ektacytometry (Lorrca MaxSis) and thoracic kyphosis angle measured in degrees on standing lateral spinal radiographs
Correlation between lumbar lordosis angle and Erythrocyte deformability (EImax) | At baseline (single time point)
  Erythrocyte deformability (EImax), measured using laser-optical ektacytometry (Lorrca MaxSis) and lumbar lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between angle of trunk rotation (ATR) and Erythrocyte deformability (EImax) | At baseline (single time point)
  Erythrocyte deformability (EImax), measured using laser-optical ektacytometry (Lorrca MaxSis) and angle of trunk rotation (ATR) measured with a scoliometer
Correlation between vertebral rotation (Nash-Moe grade) and Erythrocyte deformability (EImax) | At baseline (single time point)
  Erythrocyte deformability (EImax), measured using laser-optical ektacytometry (Lorrca MaxSis) and Vertebral rotation will be assessed using the Nash-Moe grading system on standing posteroanterior spinal radiographs. The Nash-Moe method classifies pedicle asymmetry into 5 grades (Grade 0 to Grade 4), where higher grades indicate increased vertebral rotation.
Correlation between joint hypermobility (Beighton score) and Erythrocyte deformability (EImax) | At baseline (single time point)
  Erythrocyte deformability (EImax), measured using laser-optical ektacytometry (Lorrca MaxSis) and Joint hypermobility will be measured using the Beighton score (0-9 scale), a standardized clinical examination evaluating passive dorsiflexion of the fifth finger, thumb apposition, elbow hyperextension, knee hyperextension, and forward flexion of the trunk. Scores ≥5 will be considered indicative of generalized joint hypermobility.
Correlation between Cobb angle and Erythrocyte deformability (SS1/2) | At baseline (single time point)
  Erythrocyte deformability (SS1/2), measured using laser-optical ektacytometry (Lorrca MaxSis) and Cobb angle measured in degrees on standing posteroanterior spinal radiographs
Correlation between cervical lordosis angle and Erythrocyte deformability (SS1/2) | At baseline (single time point)
  Erythrocyte deformability (SS1/2), measured using laser-optical ektacytometry (Lorrca MaxSis) and cervical lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between thoracic kyphosis angle and Erythrocyte deformability (SS1/2) | At baseline (single time point)
  Erythrocyte deformability (SS1/2), measured using laser-optical ektacytometry (Lorrca MaxSis) and thoracic kyphosis angle measured in degrees on standing lateral spinal radiographs
Correlation between lumbar lordosis angle and Erythrocyte deformability (SS1/2) | At baseline (single time point)
  Erythrocyte deformability (SS1/2), measured using laser-optical ektacytometry (Lorrca MaxSis) and lumbar lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between angle of trunk rotation (ATR) and Erythrocyte deformability (SS1/2) | At baseline (single time point)
  Erythrocyte deformability (SS1/2), measured using laser-optical ektacytometry (Lorrca MaxSis) and angle of trunk rotation (ATR) measured with a scoliometer
Correlation between vertebral rotation (Nash-Moe grade) and Erythrocyte deformability (SS1/2) | At baseline (single time point)
  Erythrocyte deformability (SS1/2), measured using laser-optical ektacytometry (Lorrca MaxSis) and Vertebral rotation will be assessed using the Nash-Moe grading system on standing posteroanterior spinal radiographs. The Nash-Moe method classifies pedicle asymmetry into 5 grades (Grade 0 to Grade 4), where higher grades indicate increased vertebral rotation.
Correlation between joint hypermobility (Beighton score) and Erythrocyte deformability (SS1/2) | At baseline (single time point)
  Erythrocyte deformability (SS1/2), measured using laser-optical ektacytometry (Lorrca MaxSis) and Joint hypermobility will be measured using the Beighton score (0-9 scale), a standardized clinical examination evaluating passive dorsiflexion of the fifth finger, thumb apposition, elbow hyperextension, knee hyperextension, and forward flexion of the trunk. Scores ≥5 will be considered indicative of generalized joint hypermobility.
Correlation between Cobb angle and Erythrocyte aggregation (AI) | At baseline (single time point)
  Erythrocyte aggregation (AI), measured using Lorrca MaxSis under standardized conditions at 37°C and Cobb angle measured in degrees on standing posteroanterior spinal radiographs
Correlation between cervical lordosis angle and Erythrocyte aggregation (AI) | At baseline (single time point)
  Erythrocyte aggregation (AI), measured using Lorrca MaxSis under standardized conditions at 37°C and cervical lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between thoracic kyphosis angle and Erythrocyte aggregation (AI) | At baseline (single time point)
  Erythrocyte aggregation (AI), measured using Lorrca MaxSis under standardized conditions at 37°C and thoracic kyphosis angle measured in degrees on standing lateral spinal radiographs
Correlation between lumbar lordosis angle and Erythrocyte aggregation (AI) | At baseline (single time point)
  Erythrocyte aggregation (AI), measured using Lorrca MaxSis under standardized conditions at 37°C and lumbar lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between angle of trunk rotation (ATR) and Erythrocyte aggregation (AI) | At baseline (single time point)
  Erythrocyte aggregation (AI), measured using Lorrca MaxSis under standardized conditions at 37°C and angle of trunk rotation (ATR) measured with a scoliometer
Correlation between vertebral rotation (Nash-Moe grade) and Erythrocyte aggregation (AI) | At baseline (single time point)
  Erythrocyte aggregation (AI), measured using Lorrca MaxSis under standardized conditions at 37°C and Vertebral rotation will be assessed using the Nash-Moe grading system on standing posteroanterior spinal radiographs. The Nash-Moe method classifies pedicle asymmetry into 5 grades (Grade 0 to Grade 4), where higher grades indicate increased vertebral rotation.
Correlation between joint hypermobility (Beighton score) and Erythrocyte aggregation (AI) | At baseline (single time point)
  Erythrocyte aggregation (AI), measured using Lorrca MaxSis under standardized conditions at 37°C and joint hypermobility (Beighton score).
Correlation between Cobb angle and Erythrocyte aggregation (Tr) | At baseline (single time point)
  Erythrocyte aggregation (Tr), measured using Lorrca MaxSis under standardized conditions at 37°C and Cobb angle measured in degrees on standing posteroanterior spinal radiographs
Correlation between cervical lordosis angle and Erythrocyte aggregation (Tr) | At baseline (single time point)
  Erythrocyte aggregation (Tr), measured using Lorrca MaxSis under standardized conditions at 37°C and cervical lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between thoracic kyphosis angle and Erythrocyte aggregation (Tr) | At baseline (single time point)
  Erythrocyte aggregation (Tr), measured using Lorrca MaxSis under standardized conditions at 37°C and thoracic kyphosis angle measured in degrees on standing lateral spinal radiographs
Correlation between lumbar lordosis angle and Erythrocyte aggregation (Tr) | At baseline (single time point)
  Erythrocyte aggregation (Tr), measured using Lorrca MaxSis under standardized conditions at 37°C and lumbar lordosis angle measured in degrees on standing lateral spinal radiographs
Correlation between angle of trunk rotation (ATR) and Erythrocyte aggregation (Tr) | At baseline (single time point)
  Erythrocyte aggregation (Tr), measured using Lorrca MaxSis under standardized conditions at 37°C and angle of trunk rotation (ATR) measured with a scoliometer
Correlation between vertebral rotation (Nash-Moe grade) and Erythrocyte aggregation (Tr) | At baseline (single time point)
  Erythrocyte aggregation (Tr), measured using Lorrca MaxSis under standardized conditions at 37°C and Vertebral rotation will be assessed using the Nash-Moe grading system on standing posteroanterior spinal radiographs. The Nash-Moe method classifies pedicle asymmetry into 5 grades (Grade 0 to Grade 4), where higher grades indicate increased vertebral rotation.
Correlation between joint hypermobility (Beighton score) and Erythrocyte aggregation (Tr) | At baseline (single time point)
  Erythrocyte aggregation (Tr), measured using Lorrca MaxSis under standardized conditions at 37°C and joint hypermobility (Beighton score)

CONTACTS AND LOCATIONS:
Overall Officials: Papatya Keles, professor, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional policies. The data contains sensitive health information that cannot be sufficiently de-identified for public distribution.

REFERENCES:
- See also: Lazari D, Freitas Leal JK, Brock R, Bosman G. The Relationship Between Aggregation and Deformability of Red Blood Cells in Health and Disease. Front Physiol 2020;11:288. — https://pmc.ncbi.nlm.nih.gov/articles/PMC7174766/
- See also: Ebenuwa I, Violet P-C, Tu H, Lee C, Munyan N, Wang Y, et al. Altered RBC deformability in diabetes: clinical characteristics and RBC pathophysiology. Cardiovasc Diabetol 2024;23:370. — https://cardiab.biomedcentral.com/articles/10.1186/s12933-024-02453-2